CLINICAL TRIAL: NCT00495287
Title: Phase III Trial in AML Comparing Standard-dose vs High-dose Remission Induction and, Within a Risk-oriented Postremission Strategy, Autologous Blood Stem Cell Transplantation vs Blood Stem Cell-supported Multicycle High-dose Program
Brief Title: A Remission Induction Therapy and Risk-oriented Postremission Strategy for Adult Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northern Italy Leukemia Group (Other)
Responsible Party: Principal Investigator, DR RENATO BASSAN, Medical Doctor, Northern Italy Leukemia Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NILG-AML 02/06
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Acute myelogenous leukemia; Adult patients; Cytogenetic risk class; Clinico-cytogenetic risk model; Risk-oriented therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Remission induction arm A is with conventional chemotherapy cycle ("ICE": idarubicin, standard-dose cytarabine, etoposide)
  Interventions: Drug: cytosine arabinoside
- B (Experimental): Remission induction therapy with high-dose cytarabine sequential regimen (HD-Ara-C, idarubicin)
  Interventions: Drug: cytosine arabinoside

INTERVENTIONS:
Drug: cytosine arabinoside — Arm A: use of standard-dose cytosine arabinoside (100 mg/m2/bd iv. on days 1-7) in association with idarubicin and etoposide.
  Arm B: use of high-dose cytosine arabinoside (1000-2000 mg/m2/bd according to age +/-65 years iv. on days 1-2 and 8-9) in association with idarubicin.
  Other Names: Aracytin; Cytarabine; Cytosar

SUMMARY:
The study was set up to assess:

1. Standard-dose versus high-dose remission induction therapy. A standard ICE chemotherapy vs sequential high-dose cytarabine, with appropriate supportive/prophylactic measures, followed by morphological, cytogenetic and molecular monitoring of remission.
2. A risk-oriented postremission therapy: HR patients will be electively submitted to allogeneic stem cell transplantation (allo-SCT), whenever possible (related/unrelated donor/cord blood; ablative/non-ablative conditioning according to national and local protocols and guidelines). Provided sufficient blood stem cells were previously collected (>2x10e6/kg Cluster of Differentiation 34 cells), SR patients and HR patients excluded from allo-SCT and aged 65 years or less will be randomized to: myeloablative autologous blood stem cell transplantation vs non-myeloablative, multicycle, autologous blood stem cell-supported high-dose cytarabine-based therapy.

   * HR/SR patients unable to be randomized because of inadequate blood stem cell yield will receive intermediate-dose consolidation; patients aged >65 years will be treated with age-adapted therapy.

DETAILED DESCRIPTION:
Adult AML is a difficult-to-treat illness because of both biological and therapeutic reasons. Most patients are aged >50 years and/or present with comorbid conditions and/or display high-risk AML-related features (poor risk, cytogenetics, prior myelodysplasia, secondary AML). This results in unsatisfactory response to conventional first-line therapy and makes it difficult to apply the most effective post-remission consolidation options (allo-SCT in younger patients with HR features, autologous blood stem cell transplantation and high-dose cytarabine-based therapy in the remainder).

In a prior, phase II uncontrolled NILG trial (registered NCT 00400637),a two-step increasing intensity induction was adopted in order to optimize induction results. 51% of ICE-refractory cases responded to the salvage regimen, irrespective of risk class. In the same study, all HR patients had to be sent to allografting whereas SR patients (by clinico-cytogenetics criteria) were to receive up to three high-dose cytarabine-based cycles, each one supported by a fixed amount of autologous blood-stem cells (1-2x10e6/kg Cluster of Differentiation 34 cells cells), to minimize the risks of high-dose cytarabine-related myelosuppression and to increase treatment intensity by reducing intercycle delays. DFS was 41% at 5 years, 58% in SR patients aged <55 years, 47% in SR patients aged >55 years, and 47% in HR patients with an identifiable donor. No treatment-related death occurred during the pancytopenic phase in 118 patients receiving 299 blood stem-cell supported high-dose cytarabine cycles.

These facts led to the present trial, in which 1) high-dose induction formerly used as salvage is directly compared to standard ICE chemotherapy and 2) the blood-stem cell supported multicycle high-dose cytarabine program is directly compared to a standard autologous blood stem cell transplantation.

RANDOM 1 CYCLE 1

* Standard ICE (all drugs by IV route): idarubicin 12 mg/m2/d on dd 1-3, cytarabine 100 mg/m2/bd on dd 1-7, etoposide 100 mg/m2/d on dd 1-5, G-CSF from d 11.
* High-dose sequential (all drugs by IV route): cytarabine 2* g/m2/bd on dd 1-2 and 8-9, idarubicin 18 mg/m2/d on dd 3 and 10, G-Colony Stimulating Factory (G-CSF) from d 11. *1 g/m2 in frail patients aged 60-65 and in all those aged >65 years.

CYCLE 2 (if CR achieved after cycle 1): Standard IC: idarubicin 10 mg/m2/d on dd 1-3, cytarabine 100 mg/m2/bd on dd 1-7, G-CSF.

CYCLE 3: Intermediate-dose cytarabine 1 g/m2/bd on dd 1-4 followed by G-CSF and by stem cell collection (1-2x10e6/kg CD34+ cells in three separate bags)

ALLO-SCT (Allogeneic Stem Cells Transplantation): All HR patients are eligible to allo-SCT as first therapeutic option. Allo-SCT procedure: any type according to local protocols/guidelines.

RANDOM 2

All SR patients and HR ones excluded from allo-SCT:

* Autologous blood stem cell transplantation after BU-CY2 regimen (Busulfan 0.8 mg/kg IV on dd -8 to -5, Cy 60 mg/kg/d on dd -4 to -3, autograft on d 0 (2-6x10e6/kg CD34+ cells) and G-CSF from d +1.
* Autologous blood stem cell supported multicycle therapy (x3, monthly) with cytarabine 2 g/m2/bd on dd 1-5, idarubicin 8 mg/m2/d on dd 1-2, autograft on d 6 (1-2x10e6/kg CD34+ cells) and G-CSF from d 8.

Patients excluded from Random 2 as well as from allo-SCT receive attenuated, unsupported consolidation with 1-2 intermediate-dose cytarabine cycles. Patients aged >65 years are excluded from Random 2.

RISK CLASSIFICATION Cytogenetic risk classification is based on MRC/ECOG-SWOG/CALGB criteria (cytogenetic risk classes: favorable, normal/intermediate, unfavorable, other, unknown); clinical risk classification is based on selected diagnostic criteria and response to chemotherapy cycle 1. The final risk model integrates cytogenetic and clinical risk to encompass two broad risk classes (SR and HR).

* Standard risk (SR): favorable cytogenetics, CR achieved after cycle 1; or normal/intermediate cytogenetics, CR achieved after cycle 1, lack of high-risk characteristics.
* High risk (HR): unfavorable cytogenetics; or normal/intermediate cytogenetics with any high-risk characteristic (WBC >50x10e9/l,FAB M0,6,7 or corresponding WHO, secondary AML, Myelodysplastic Syndrome (MDS)-associated AML, hepatosplenomegaly, FLT3 mutation, CR) not achieved with cycle, persistent cytogenetic abnormality at CR), or other/unknown cytogenetics.

ELIGIBILITY:
Inclusion criteria (Random 1):

* Age 16+ years
* Diagnosis of untreated (or only hydroxyurea/cyclophosphamide) acute myelogenous leukemia (AML, including myeloid sarcoma) or high-risk myelodysplasia (RAEB-2), either de novo or following an antecedent hematological disorder, or secondary to chemo-radiotherapy for other cancer
* Signed informed consent
* Adequate sampling for full cytological, cytochemical, cytogenetic and immunobiological disease characterization by revised FAB, EGIL and WHO criteria
* ECOG performance status 0-2 or reversible ECOG 3 score following intensive care of complications.

Exclusion criteria:

* Diagnosis of acute promyelocytic leukemia
* Pre-existing, uncontrolled pathology such as cardiac disease (congestive/ischemic, acute myocardial infarction within the past 3 months, untreatable arrythmias, NYHA classes III and IV), severe liver disease with serum bilirubin >3 mg/dL and/or ALT >3 x upper normal limit (unless attributable to AML), kidney function impairment with serum creatinine >2 mg/dL (unless attributable to AML), and severe neuropsychiatric disorder that impairs the patient's ability to understand and sign the informed consent, or to cope with the intended treatment plan
* Known HIV positive serology
* Other active hematological or non-hematological cancers with life expectancy <1 year
* Pregnancy (fertile women will be advised not to become pregnant while on treatment; and male patients to adopt contraceptive methods)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2006-11; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Remission induction (R1): Complete remission (CR) rate after cycle 1 | 30 days after beginning chemotherapy.
Remission consolidation (R2): Length of remission (DFS, disease-free survival) | 5 years

SECONDARY OUTCOMES:
R1: CR with incomplete hematological recovery | 30 days after beginning chemotherapy
R1:Complete cytogenetic remission | 30 days after beginning chemotherapy
R1: Treatment-related death (TRD) | 2 months
R2: Overall survival (OS) | 5 years
Remission duration and cumulative incidence of relapse | 5 years
Treatment-related death | 5 years
Quality of Life | 1 year and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Renato Bassan, MD, Principal Investigator — Norther Italy Leukemia Group
Locations (17):
- Italy (17):
  - Dipartimento di Ematologia e Medicina Trasfusionale - Azienda Osp. Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - USC Ematologia Azienda Papa Giovanni XXIII, Bergamo, BG
  - Ospedale Spedali Civili di Brescia, Brescia, Brescia
  - Ospedale Generale di Bolzano, Bolzano, Bz
  - S.C. Ematologia - Azienda Ospedaliera S.Croce e Carle, Cuneo, CN
  - Istituti Ospitalieri, Cremona, Cremona
  - Ematologia - AOU Careggi, Florence, FI
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ematologia Centro TMO - Fondazione IRCSS Ospedale Maggiore, Milan, MI
  - Ematologia e TMO - Ospedale San Raffaele, Milan, MI
  - Istituto Nazionale Dei Tumori, Milan, MI
  - Ematologia - TMO - Ospedale San Gerardo, Monza, MI
  - A.O.U San Giovanni Battista-Divisione Ematologica dell'Università, Torino, TO
  - Ematologia 2 - Osp. Molinette San Giovanni Battista, Torino, TO
  - Ospedale Mauriziano, Torino, TO
  - Ospedale di Circolo di Varese, Varese, Varese
  - Ospedale dell'Angelo, Mestre, Venezia

REFERENCES:
- [Derived] Caprioli C, Lussana F, Salmoiraghi S, Cavagna R, Buklijas K, Elidi L, Zanghi' P, Michelato A, Delaini F, Oldani E, Intermesoli T, Grassi A, Gianfaldoni G, Mannelli F, Ferrero D, Audisio E, Terruzzi E, De Paoli L, Cattaneo C, Borlenghi E, Cavattoni I, Tajana M, Scattolin AM, Mattei D, Corradini P, Campiotti L, Ciceri F, Bernardi M, Todisco E, Cortelezzi A, Falini B, Pavoni C, Bassan R, Spinelli O, Rambaldi A. Clinical significance of chromatin-spliceosome acute myeloid leukemia: a report from the Northern Italy Leukemia Group (NILG) randomized trial 02/06. Haematologica. 2021 Oct 1;106(10):2578-2587. doi: 10.3324/haematol.2020.252825. PMID 32855275
- [Derived] Gianfaldoni G, Mannelli F, Intermesoli T, Bencini S, Giupponi D, Farina G, Cutini I, Bonetti MI, Masciulli A, Audisio E, Ferrero D, Pavoni C, Scattolin AM, Bosi A, Rambaldi A, Bassan R. Early peripheral clearance of leukemia-associated immunophenotypes in AML: centralized analysis of a randomized trial. Blood Adv. 2020 Jan 28;4(2):301-311. doi: 10.1182/bloodadvances.2019000406. PMID 31978214
- [Derived] Bassan R, Intermesoli T, Masciulli A, Pavoni C, Boschini C, Gianfaldoni G, Marmont F, Cavattoni I, Mattei D, Terruzzi E, De Paoli L, Cattaneo C, Borlenghi E, Ciceri F, Bernardi M, Scattolin AM, Todisco E, Campiotti L, Corradini P, Cortelezzi A, Ferrero D, Zanghi P, Oldani E, Spinelli O, Audisio E, Cortelazzo S, Bosi A, Falini B, Pogliani EM, Rambaldi A. Randomized trial comparing standard vs sequential high-dose chemotherapy for inducing early CR in adult AML. Blood Adv. 2019 Apr 9;3(7):1103-1117. doi: 10.1182/bloodadvances.2018026625. PMID 30948365